CLINICAL TRIAL: NCT03133624
Title: This is a Registry Study on a Multidimensional Prediction Model for Rupture Risk of Unruptured Intracranial Aneurysms in China
Brief Title: A Study on a Multidimensional Prediction Model for Rupture Risk of Unruptured Intracranial Aneurysms
Acronym: CIAP-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Xinjian Yang, MD, Vice Chair of Department of Interventional Neuroradiology of Beijing Neurosurgical Institute, Beijing Neurosurgical Institute
Other Study IDs: 2016YFC1300802
Record Dates: First submitted 2017-04-16; First posted 2017-04-28 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Intracranial Aneurysm
Keywords: unruptured intracranial aneurysms; rupture risk; computational fluid dynamic; high resolution magnetic resonance images; gene; multi dimensional prediction model; clinical features; risk factors; registry study; china; biomarkers
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a registry study on a multidimensional prediction model for rupture risk of unruptured intracranial aneurysms in China.

DETAILED DESCRIPTION:
This subsequent program China Intracranial Aneurysm Project - 2 (CIAP-2) will comprise screening of 500 patients from the UIA cohort (CIAP-1) and focus on hemodynamics factors, high resolution magnetic resonance imaging (HRMRI), genetic factors and biomarkers. Possible risk factors for rupture of UIA, including genetic factors, biomarkers, HRMRI, and hemodynamic will be analyzed. The first project of the China Intracranial Aneurysm Project (CIAP-1: Chaired by the Department of Neurosurgery, Tangdu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China) will establish a prospective cohort of 5000 patients with UIA from 20 centers in China, and collect baseline information for each patient. Multidimensional data will be acquired in follow-up assessments. Statistically significant clinical features in the UIA cohort will also be analyzed and integrated into this model for predicting risk of UIA rupture. After the model has been set up, the resultant evidence-based prediction will be used to provide a preliminary theoretical basis for the treatment of aneurysms at high risk of rupture.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 UIA that is untreated and confirmed by imaging: Computed tomography angiography (CTA), magnetic resonance angiography (MRA) and digital subtraction angiography (DSA). Regardless of the presence of clinical symptoms
* Patient currently has the ability to live independently, and a modified Ranking Score less than or equal to 3 points
* Older than 14 years of age
* Patient or relatives agreed to sign the consent form

Exclusion Criteria:

* Subarachnoid hemorrhage of unknown origin
* Presence of other intracranial vascular malformations, such as cerebral arteriovenous malformation (AVM) or cerebral arteriovenous fistula (AVF)
* Intracranial and other malignant tumors
* Fusiform, traumatic, bacterial or dissecting aneurysm
* Patients with severe mental illness who are unable to communicate
* Patients with other diseases or poor general condition who are expected to survive less than 1 year
* Patients with intracranial aneurysms who have joined other similar research institutions
* Patients who refused follow-up

The definition of modified Ranking Score:

* 0 Completely silent
* 1 Despite symptoms, but not visibly disabled, can complete all regular duties and activities
* 2 Mild disabilities, not all activities previously possible, but can deal with personal affairs without need of assistance
* 3 Moderate disability requires some help, but walking does not need assistance;
* 4 Severe disabilities, unable to walk independently, no others can not meet their needs
* 5 Severely disabled, bedridden, Urine, requiring continuous care and care;
* 6 Mortality

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with at least 1 UIA that is untreated and confirmed by imaging (CTA, MRA and DSA), regardless of the presence of clinical symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The rupture of intracranial aneurysms | Up to 12 months or time of aneurysm repair surgery
  The rupture of unruptured intracranial aneurysms.

SECONDARY OUTCOMES:
Changes in morphology of unruptured intracranial aneurysms | Up to 12 months or time of aneurysm repair surgery
  Maximum diameter increase ≥ 1mm or appearance of a daughter sac.

CONTACTS AND LOCATIONS:
Overall Officials: Xinjian Yang, MD, Principal Investigator — Beijing Neurosurgical Institute and Beijing Tiantan Hospital affiliated to Capital Medical University，China
Locations (12):
- China (12):
  - XuanWu Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The 1st Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Southern Medical University, Zhujiang Hospital, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Liao Cheng People's Hospital, Liaocheng, Shandong
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Neurosurgery, Tangdu Hospital, Fourth Military Medical University Xi'an, China, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital Of Xinjiang Medical University, Ürümqi, Xinjiang
  - Beijing Neurosurgical Institute and Beijing Tiantan Hospital affiliated to Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
we can share the original data 5 years after the study.

REFERENCES:
- [Result] International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms--risk of rupture and risks of surgical intervention. N Engl J Med. 1998 Dec 10;339(24):1725-33. doi: 10.1056/NEJM199812103392401. PMID 9867550
- [Result] UCAS Japan Investigators; Morita A, Kirino T, Hashi K, Aoki N, Fukuhara S, Hashimoto N, Nakayama T, Sakai M, Teramoto A, Tominari S, Yoshimoto T. The natural course of unruptured cerebral aneurysms in a Japanese cohort. N Engl J Med. 2012 Jun 28;366(26):2474-82. doi: 10.1056/NEJMoa1113260. PMID 22738097
- [Result] Thompson BG, Brown RD Jr, Amin-Hanjani S, Broderick JP, Cockroft KM, Connolly ES Jr, Duckwiler GR, Harris CC, Howard VJ, Johnston SC, Meyers PM, Molyneux A, Ogilvy CS, Ringer AJ, Torner J; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention; American Heart Association; American Stroke Association. Guidelines for the Management of Patients With Unruptured Intracranial Aneurysms: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Aug;46(8):2368-400. doi: 10.1161/STR.0000000000000070. Epub 2015 Jun 18. PMID 26089327
- [Result] Liu J, Xiang J, Zhang Y, Wang Y, Li H, Meng H, Yang X. Morphologic and hemodynamic analysis of paraclinoid aneurysms: ruptured versus unruptured. J Neurointerv Surg. 2014 Nov;6(9):658-63. doi: 10.1136/neurintsurg-2013-010946. Epub 2013 Nov 12. PMID 24220206
- [Result] Li MH, Chen SW, Li YD, Chen YC, Cheng YS, Hu DJ, Tan HQ, Wu Q, Wang W, Sun ZK, Wei XE, Zhang JY, Qiao RH, Zong WH, Zhang Y, Lou W, Chen ZY, Zhu Y, Peng DR, Ding SX, Xu XF, Hou XH, Jia WP. Prevalence of unruptured cerebral aneurysms in Chinese adults aged 35 to 75 years: a cross-sectional study. Ann Intern Med. 2013 Oct 15;159(8):514-21. doi: 10.7326/0003-4819-159-8-201310150-00004. PMID 24126645
- [Derived] Fan XX, Geng JW, He C, Hu P, Sun LY, Zhang HQ. Analysis of the wall thickness of intracranial aneurysms: Can computational fluid dynamics detect the translucent areas of saccular intracranial aneurysms and predict the rupture risk preoperatively? Front Neurol. 2023 Jan 9;13:1075078. doi: 10.3389/fneur.2022.1075078. eCollection 2022. PMID 36698880
- [Derived] Chen J, Liu J, Zhang Y, Tian Z, Wang K, Zhang Y, Mu S, Lv M, Jiang P, Duan C, Zhang H, Qu Y, He M, Yang X. China Intracranial Aneurysm Project (CIAP): protocol for a registry study on a multidimensional prediction model for rupture risk of unruptured intracranial aneurysms. J Transl Med. 2018 Sep 26;16(1):263. doi: 10.1186/s12967-018-1641-1. PMID 30257699